CLINICAL TRIAL: NCT04625855
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr) Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Study of the Absorption, Metabolism, and Excretion of [14C]-Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr) Following a Single Oral Dose in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPR994-106
Record Dates: First submitted 2020-09-17; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Healthy Volunteers
Keywords: pharmacokinetics; TBPM-PI-HBr; tebipenem; absorption; metabolism; excretion

STUDY DESIGN:
Intervention Model Description: Single-Center, Open-Label, Non-Randomized, Phase 1 Study
Masking Description: None (Open-Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TBPM-PI-HBr (Experimental): Healthy subjects meeting eligibility criteria will receive a single dose of 600mg of TBPM-PI-HBr
  Interventions: Drug: TBPM-PI-HBr

INTERVENTIONS:
Drug: TBPM-PI-HBr — TBPM-PI-HBr (3 x 200 mg tablets) once
  Other Names: TBPM-PI-HBr oral capsule

SUMMARY:
The purpose of this study is to determine the absorption, metabolism, and excretion of [14C]-TBPM-PI-HBr and to characterize and determine the metabolites present in plasma, urine, and where possible, feces in healthy male subjects following a single oral administration.

ELIGIBILITY:
Inclusion Criteria

* Healthy adult males, of any race, between 18 and 55 years of age, inclusive.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive, and a total body weight between 50 and 100 kg, inclusive at Screening.
* Willing and able to provide written informed consent and comply with all study assessments, restrictions, and adhere to the protocol schedule.
* Medically healthy with no clinically significant medical history, or abnormalities in physical examination, laboratory variables, vital signs or ECG at the time of screening and Check-in, as deemed by the Investigator (or designee).
* Have suitable venous access for repeated blood sampling.
* History of a minimum of 1 bowel movement per day.

Exclusion Criteria

* History or suspicion of routine or chronic drug or alcohol abuse or dependence within 2 years prior to Check-in.
* Use of tobacco, nicotine, or nicotine-replacement products within 30 days prior to Check-in or planned use during the study.
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
* Use/receipt of any prescription or nonprescription medication, herbal products, vitamins or vaccines within 14 days (or 5 half-lives whichever is longer) prior to Check-in, without prior approval from the Medical Monitor.
* Donation of more than 500 mL of blood or plasma within 56 days prior to Check-in, or receipt of a blood transfusion within 1 year prior to Check-in.
* Receipt of any other investigational product or participation in another investigational clinical study that included drug treatment within 30 days, or 5 times the t1/2 of the investigational drug, whichever is longer.
* Have previously completed or withdrawn from this study or any other study investigating TBPM-PI-HBr, and have previously received TBPM-PI-HBr.
* Subjects with exposure to significant diagnostic or therapeutic radiation (e.g., serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in.
* Subjects who have participated in a radiolabeled drug study where exposures are known to the Investigator within the previous 3 months prior to admission to the clinic for this study or participated in a radiolabeled drug study where exposures are not known to the Investigator within the previous 6 months prior to admission to the clinic for this study. The total 12-month exposure from this study and a maximum of 3 other previous radiolabeled studies within 3 to 12 months prior to this study will be within the CFR recommended levels considered safe, per United States (US) Title 21 CFR 361.1.
* Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy adult males, of any race
Enrollment: 8 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of Tebipenem (TBPM) will be determined following administration of [14C]-TBPM-PI-HBr to healthy male subjects | Day 1 to Day 5
  The primary PK outcome endpoints following oral administration of [14C]-TBPM-PI-HBr will be derived for TBPM in plasma (calculated from whole blood concentrations) based on the concentration-time profile
Total radioactivity will be determined following administration of [14C]-TBPM-PI-HBr to healthy male subjects | Day 1 to Day 5
  The primary PK outcome endpoints following oral administration of [14C]-TBPM-PI-HBr will be derived for total radioactivity in whole blood and plasma based on the total radioactivity concentration-time profile

SECONDARY OUTCOMES:
Metabolite profiling and chemical structuring of metabolites in plasma, urine, and, where possible, feces will be determined after a single oral dose of [14C]-TBPM-PI-HBr | Day 1 to Day 5
  The secondary metabolite outcome endpoints will be derived:
  * metabolic profile of TBPM-PI-HBr
  * metabolic profile of TBPM-PI-HBr
Metabolite profiling and chemical structuring of metabolites in plasma, urine, and, where possible, feces will be determined after a single oral dose of [14C]-TBPM-PI-HBr | Day 1 to Day 5
  The secondary metabolite outcome endpoints will be derived:
  • identification of the structure of TBPM-PI-HBr metabolites
The safety and tolerability of a single oral dose of [14C]-TBPM-PI-HBr when administered to healthy male subjects. | Day 1 to Day 5
  The secondary safety outcome measures for this study are as follows:
  • incidence and severity of AEs
The safety and tolerability of a single oral dose of [14C]-TBPM-PI-HBr when administered to healthy male subjects. | Day 1 to Day 5
  The secondary safety outcome measures for this study are as follows:
  •incidence of laboratory abnormalities, based on hematology, clinical chemistry, coagulation, and urinalysis test results

CONTACTS AND LOCATIONS:
Overall Officials: Irene Mirkin, MD, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No